CLINICAL TRIAL: NCT02349243
Title: Effect of Entacapone on Bodyweight Loss in Obese Population: A Randomized, Double-blind, Placebo-controlled, Pilot Trial
Brief Title: Effect of Entacapone on Bodyweight Loss in Obese Population
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaichun Wu (Other)
Collaborators: National Institute of Biological Sciences, Beijing (Unknown)
Responsible Party: Sponsor-Investigator, Kaichun Wu, Dr., Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJETKP01
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Obesity
Keywords: obese; weight loss; entacapone
MeSH Terms: conditions — Obesity; Weight Loss | interventions — entacapone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- entacapone (Experimental): An approach of 200mg entacapone at a time and 4 times a day(0.5 hour after every breakfast, lunch and supper and at 0.5 hours before bedtime) is adopted. Every participant is required to record his/her diet, exercise, and drug intake condition in a standard record card which is provided by the researchers.
  Interventions: Drug: Entacapone
- placebo (Placebo Comparator): Except for taking the placebo rather than the entacapone, any intervention in the placebo group is the same with that in the entacapone group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Entacapone — 200 mg entacapone, oral intake, 4 times per day (after breakfast, lunch, supper and before sleep at night), for 6 six months
  Other Names: Comtan
  Arms: entacapone
Drug: Placebo — 200 mg placebo, oral intake, 4 times per day (after breakfast, lunch, supper and before sleep at night), for 6 six months
  Other Names: Sugar pills manufactured to mimic entacapone 200mg tablet
  Arms: placebo

SUMMARY:
This is a randomized, controlled, double blind clinical trial. The purpose of this study is to investigate the weight loss efficacy of entacapone. In this study, participants are randomly divided into entacapone and placebo groups. The percentage change in body weight, the body mass index, waist circumstance, extent of fatty liver, quantity of visceral fat, serum insulin, serum triglyceride and the adverse effects are compared between the two groups.

DETAILED DESCRIPTION:
All volunteers should clearly understand the objectives and the risks of the present study. Then, all volunteers should carefully read and sign the informed consent and receive a copy of the signed informed consent. If the volunteer agrees to participate to the present study and signs the informed consent, the volunteer is included. The included participants should be followed up and the case report form should be competed by appointed researchers.

Recruiting stage:

To check whether a volunteer are eligible to participate:

1. All volunteers are checked according to the inclusive and the exclusive criteria;
2. The clinical nutritionists provide diet and exercise regime to the volunteers.

Grouping stage:

A group of 12 Participants enter the study at a time,

1. To assess the performance of the volunteer complying the diet and exercise regime;
2. Volunteers who are able to comply the regime and sign the informed consent are included;
3. Every participate receives a random number which is packed in an opaque envelop;
4. Physical examination: blood pressure, heart rate, height, bodyweight, waist and hip circumference;
5. Laboratory examination: level of adiponectin, leptin, resistin, C-reactive protin, insulin, fasting blood glucose, haemoglobin A1c, tri glycerides, total cholesterol, LDL cholesterol, HDL cholesterol;
6. Extra blood sample(20ml) is collected to measure the level of adiponectin, resistin and leptin;
7. The opaque envelop contained the random number is opened by the CRA and the grouping is determined;
8. Participants take entacapone or placebo as the physicians and researchers have instructed and make a record in a standard form;
9. Participants carry out the diet and exercise regime, measure their bodyweight everyday and take a record.

Intervening stage:

1. Two weeks after the first intervention, monthly telephone interview start:

   1.1 Ask the participant the details of taking medicine, following the diet and exercise regime, the present body weight; 1.2 Ask the participant whether they have any discomfort and to decide whether medical interventions are needed.
2. Four weeks after the first intervention, monthly hospital interview start:

2.1 The day before the participants go to hospital for the second interview. 2.1.1 Any drink, food and strenuous activity should be avoided at least 8 hours before the second interview; 2.1.2 The standard form of daily activity should be brought. 2.2 During this interview: 2.2.1 Physical examination：blood pressure, heart rate, height, bodyweight, waist and hip circumference; 2.2.2 The details of participants taking medicine, following the diet and exercise regime should be asked; 2.2.3 Laboratory examination: level of adiponectin, leptin, resistin, C-reactive protin, insulin, fasting blood glucose, haemoglobin A1c, triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol; 2.2.4 20ml blood sample is collected to measure the level of adiponectin, resistin, leptin and the expression of obese related genes; 2.2.5 Abdominal MRI should be made; 2.2.6 Any discomfort of the participants should be recorded and medical treatment should be provided when it is necessary; 2.2.7 The previous standard form of daily activity are hand over to the CRA and blank forms are provided; 2.2.8 The untaken drugs should be retrieved, packed and a record should be maed; 2.2.9 Drugs of the next month should be distributed and a relevant record should be made.

2.3 Participate go back home. 2.3.1 Participants continue to take entacapone or placebo as the physicians and researchers have instructed and make a record in a standard form; 2.3.2 Participants continue to carry out the diet and exercise regime, measure their bodyweight everyday and take a record.

All the data should be recorded in a standard case report form and the accuracy, completeness and timeliness be regularly checked by an appointed clinical research associate.

The sample size is calculated by the software PASS 11.0. The alternative hypothesis set as Mean 1<Mean 2, which means that the participants in the entacapone group loss more weight than the participants in the placebo group. Because this is a pilot study, the error is set as (1-β)=0.8 and α=0.1. According to the results of the study on tesofensine, another weight loss drug, participants in the entacapone and placebo group are estimated to loss 2 kg and 10 kg respectively. The estimated sample size is 30, 15 in each arm.

The statistical analysis is conducted by the computer software SPSS 17.0.0 (SPSS Inc, Chicago, Ill). All analyses are performed according to the intention-to-treat principle. The occurrences of the primary and secondary end points are compared between the entacapone and placebo groups. The categorical data are reported as numbers with proportions, and the quantitative data are reported as medians with interquartile ranges (IQRs) or means with standard deviation. The categorical data were compared using the Chi-squared or Fisher exact test where appropriate. For the continuous data, the Mann-Whitney U-test were used for the group comparisons as appropriate. A two-sided p value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1) Obese which is defined as BMI ≥ 28kg/m2 ;
* 2) 18≤ age ≤60 years;
* 3) Permanent resident in Xi'an City, Shaanxi Province, China

Exclusion Criteria:

* 1) Unable to closely follow the diet and exercise regime;
* 2) Bodyweight changes beyond 4kg within 3 month before participating in this study;
* 3) Have a history of myocardial infarction or unstable angina within 6 month before participating in this study;
* 4) With endocrine, neurological, psychiatric or malignant diseases;
* 5) History of thyroid diseases;
* 6) Cardiac, hepatic and renal dysfunction;
* 7) Have a long history of using amcinonide;
* 8) With intestinal malabsorption;
* 9) With history of acute or chronic pancreatitis
* 10) With history of gastrointestinal surgery;
* 11) With history of bariatric surgery;
* 12) Using any other pharmacological drugs for weight loss;
* 13) Addicted to any drugs including alcohol;
* 14) Diabetes;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Percentage change in bodyweight | Monthly until the 6th month after the 1st intervention
  The final result will be assessed six months after intervention

SECONDARY OUTCOMES:
Changes in body mass index | Monthly until the 6th month after the 1st intervention
Waist circumstance | Monthly until the 6th month after the 1st intervention
Visceral adipose tissue | Monthly until the 6th month after the 1st intervention
Serum adipokines | Monthly until the 6th month after the 1st intervention
  level of adiponectin, leptin, resistin, C-reactive protein
glucose tolerance index | Monthly until the 6th month after the 1st intervention
  insulin, fasting blood glucose, haemoglobin A1c
Dyslipidemia index | Monthly until the 6th month after the 1st intervention
  triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol
Adverse effects | Monthly until the 6th month after the 1st intervention
  pain, fatigue, back pain, sweating increased, dyskinesias, dizziness, nausea, diarrhea, abdominal pain, constipation, mouth dry, hallucination, upper respiratory tract infection, fall, urine abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, MD, PhD, Study Chair — Xijing Hospital of Digestive Diseases, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China